CLINICAL TRIAL: NCT04602494
Title: Varenicline For Nicotine Vaping Cessation In Non Smoker Vaper Adolescents
Acronym: Pilot
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The pilot study used apo-varenicline under temp FDA authorization. When varenicline was available an IND exemption was granted to enroll children, IRB approved a trial of varenicline in participants ages 16-25 June 27, 2022, the pilot was terminated
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, A. Eden Evins, Founder Director, Center for Addiction Medicine and Director for Faculty Development, Department of Psychiatry; Cox Family Professor of Psychiatry in the Field of Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P002774-Pilot; R01DA052583 (NIH)
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Vaping; Nicotine Dependence
Keywords: Vaping; Nicotine; Adolescents; Cessation; Varenicline
MeSH Terms: conditions — Vaping; Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: This a 3-arm, randomized, placebo-controlled, parallel-group design of (1) varenicline up to 1 mg bid for 12 weeks added to behavioral and texting support vaping cessation compared or (2) behavioral and texting support and placebo or (3) monitoring only.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomly assigned in a 1:1:1 ratio, in blocks of 6, to double-blind varenicline, identical placebo prepared by the MGH research pharmacy or monitoring (i.e., assessment only). Randomization will be computer generated by the MGH Research Pharmacy personnel with no other interactions with study staff or participants. The full randomization code (drug, placebo, monitoring) will be held in the MGH research pharmacy and available to study PI only in the case of urgent medical need. A partial randomization code (treatment vs monitoring) will be held by the interventionist at the Center for Addiction Medicine. Participants, investigators and outcome assessor will remain fully blind to all 3 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Varenicline (Experimental): Participants will receive varenicline 0.5 mg once daily on days 1-3, 0.5 mg twice daily on days 4-7 and starting on day 8, 1 mg twice daily for a total of 12 weeks added to 12 weeks of group behavioral and texting support specifically designed for teen vaping cessation
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Participants will receive identical placebo 0.5 mg once daily on days 1-3, 0.5 mg twice daily on days 4-7 and starting on day 8, 1 mg twice daily for a total of 12 weeks added to 12 weeks of group behavioral and texting support specifically designed for teen vaping cessation
  Interventions: Drug: Placebo
- Monitoring only (No Intervention): Participants will attend weekly and monthly sessions that will only consist of assessments. No study medication, no behavioral or texting support.

INTERVENTIONS:
Drug: Varenicline — varenicline: 0.5 mg once daily on days 1-3, 0.5 mg twice daily on days 4-7 and starting on day 8, 1 mg twice daily for a total of 12 weeks
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Identical placebo: 0.5 mg once daily on days 1-3, 0.5 mg twice daily on days 4-7 and starting on day 8, 1 mg twice daily for a total of 12 weeks
  Arms: Placebo

SUMMARY:
The Investigators propose a randomized, placebo-controlled trial to test the hypothesis that varenicline added to group behavioral and texting support will be well tolerated and improve vaping cessation rates among nicotine dependent adolescents who vape, do not smoke regularly, and are willing to try treatment to stop vaping compared to placebo added to group behavioral and texting support. The study will consist of a three-arm randomized, placebo-controlled, parallel-group study of (1) varenicline up to 1 mg bid for 12 weeks added to behavioral and texting support compared with (2) behavioral and texting support and placebo and (3) monitoring only. The primary comparison will be of vaping cessation rates in those assigned to varenicline vs placebo.To do this, the investigators propose to enroll 300 adolescents aged 16-25 who meet eligibility criteria.

DETAILED DESCRIPTION:
Enrollees will include 300 nicotine dependent adolescents aged 16-25, who vape, do not smoke, and want to quit vaping. The study will will consist of a three-arm randomized, placebo-controlled, parallel-group study of (1) varenicline up to 1 mg bid for 12 weeks added to behavioral and texting support for adolescent vaping cessation or (2) behavioral and texting support and placebo or (3) monitoring only. The primary comparison of interest is efficacy of (1) varenicline vs (2) placebo arms on vaping abstinence outcomes. The study consists of one enrollment visit, one baseline visit, twelve weekly individual treatment and assessment sessions, and six monthly visits at weeks 4, 8, 12, 16, 20 and 24 weeks. At the enrollment visit, participants will complete interviews, questionnaires and diagnostic assessments, as well as saliva and urine sample and vitals. At the baseline visit, participants will complete several interviews, questionnaires, provide a saliva sample for cotinine measurement, and be randomized to the varenicline plus behavioral treatment group, the placebo plus behavioral treatment group, or monitoring-only group. Study staff will distribute varenicline or identically appearing placebo with instructions on how to take the study medication at weeks 0, 2, 4 and 8. Participants will be instructed to bring all empty and unused study medication at each in-person study visit through Week 12. At the weekly treatment meetings, participants will participate in cognitive behavioral therapy and complete questionnaires. Monthly visits will consist of interviews, questionnaires and a saliva and urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-25 inclusive;
* Self report of daily or near daily nicotine vaping for the prior ≥ 3 months, screening semi-quantitative urine cotinine positive for recent nicotine use, exhaled CO <10 ppm and score ≥4 on the 10-item E-cigarette Dependence Inventory (ECDI);
* Self-report of no combusted tobacco use in the past 2 months at enrollment;
* Total body weight at screening ≥35 kg (77 lbs) and Body Mass Index (BMI) ≤35 kg/m2;
* Report motivation to quit vaping in the next 30 days;
* Able to understand study procedures and read and write in English;
* Competent and willing to consent to participate in study procedures.

Exclusion Criteria:

* Use of a smoking cessation medication in the prior month (nicotine patch, gum, nasal spray, or inhaler, varenicline, bupropion);
* Unwillingness to abstain during the study from using smoking cessation aids other than those provided by the study;
* Unstable medical condition, epilepsy, severe renal impairment;
* Evidence of active problem substance use severe enough in the investigator's opinion to compromise ability to safely participate;
* Prior adverse drug reaction to varenicline;
* Unwilling to provide urine samples;
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eden Evins, MD, Principal Investigator — Massachusetts General Hospital; Randi Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Addiction Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices), and the study protocol, statistical analysis plan, analytic code, and informed consent form will be made available to researchers who provide a methodologically sound proposal beginning 3 months and ending 5 years following article publication to achieve aims in the approved proposal. Proposals should be directed to rschuster@mgh.harvard.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Data access agreement required.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five participants signed consent and were enrolled. One (1) subject was considered a screen fail and not randomized to an arm/group, and four (4) subjects were randomized.
Period: Overall Study
Arm/Group | Varenicline | Placebo | Monitoring Only
Started | 1 | 1 | 2
Completed | 1 | 1 | 0
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Monitoring Only | Total
Number analyzed (Participants) | 1 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (0) | 21 (0) | 21.5 (0.50) | 21.25 (0.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 1 | 2 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Continuous Nicotine Vaping Abstinence From Week 9 Through End of Treatment (Week 12)
Description: Those assigned to varenicline and group behavioral and texting support will have a higher rate of cotinine verified, continuous nicotine vaping abstinence from study week 9 to end of treatment as operationalized by self-report of no nicotine vaping since the last study visit on a timeline followback assessment and urinary cotinine <50 ng/mL at each study visit in the designated timeframe.
Time Frame: Weeks 9-12
Population: 5 people enrolled in the pilot, 1 was a screen fail, 4 were enrolled and have been included in the analysis. Due to the small number of participants enrolled in the pilot, data is presented as participant count.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 2
Participants | 0 | 1 | 0

2. Primary Outcome: Percentage of Participants With Continuous Nicotine Vaping Abstinence From Week 9 Through End of Follow-up (Week 24)
Description: Those assigned to varenicline and group behavioral and texting support will have a higher rate of cotinine verified, continuous nicotine vaping abstinence from study week 9 to end of follow-up as operationalized by self-report of no nicotine vaping since the last study visit on a timeline followback assessment and urinary cotinine <50 ng/ml at each study visit in the designated timeframe.
Time Frame: Weeks 9-24
Population: No participant reached 24 weeks in the study, and as such, were not included in the analysis.
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Percentage of Change in Nicotine Product Exposure
Description: Those assigned to varenicline will have greater percentage reduction in vaped nicotine product exposure than those assigned to placebo as determined by urine cotinine from baseline to week 24. Cotinine is a byproduct of nicotine that is used to measure exposure to nicotine product exposure. Positive values represent increases and negative values represent decreases.
Time Frame: Baseline-week 24
Measure: Number; unit: percentage change in nicotine exposure
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 2
percentage change in nicotine exposure | -99 | -100 | 0

4. Primary Outcome: Onset of Vaping Abstinence in Weeks
Description: Those assigned to varenicline will have earlier onset of abstinence. Onset of vaping abstinence (weeks) was assessed by participant self-report of vaping abstinence, and verified by urine cotinine testing.
Time Frame: Baseline-24 weeks
Population: No participants in the monitoring only group quit vaping.
Measure: Number; unit: Weeks
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
Weeks | 8 | 2 |

5. Primary Outcome: Latency to First Lapse in Weeks
Description: Those assigned to varenicline will have longer latency to first lapse. This outcome was assessed via self-report and verified by urine cotinine testing.
Time Frame: Baseline-24 weeks
Population: No participants in the monitoring only group quit vaping, and as such, could not lapse.
Measure: Number; unit: Weeks
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
Weeks | 10 | NA — Participant did not have a lapse from week 2 to the end of the trial. |

6. Primary Outcome: Latency to Relapse in Weeks
Description: Those assigned to varenicline will have longer latency to relapse. This outcome was assessed by self-report and verified by urine cotinine testing at each study visit.
Time Frame: Baseline-24 weeks
Population: No participants in the monitoring only group quit vaping, and as such, could not relapse.
Measure: Number; unit: Weeks
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
Weeks | NA — Participant in the varenicline group quit vaping at week 8, had a lapse at week 10, and then stayed abstinent until the end of the trial. No relapse reported. | NA — Participant in the placebo group quit vaping at week 2 and stayed abstinent until the end of the trial. No relapse reported. |

7. Primary Outcome: Duration of Vaping Abstinence in Weeks
Description: Those assigned to varenicline will have a longer duration of abstinence in weeks. This measure was assessed by self-report and verified by urine cotinine testing at each study visit.
Time Frame: Baseline-24 weeks
Population: No participants in the monitoring group quit vaping.
Measure: Number; unit: Weeks
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
Weeks | 15 | 22 |

8. Primary Outcome: Total Number of Days of Vaping Abstinence
Description: Those assigned to varenicline will have greater total number of days of vaping abstinence. Total number of days of vaping abstinence was assessed by self-report and verified by urine cotinine testing at each study visit.
Time Frame: Baseline-24 weeks
Population: No participant reached 24 weeks in the study, and as such, were not included in the analysis.
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Adverse Events During the Treatment Period
Description: Adverse events are assessed via standardized questions prompting participants to report any changes in their physical or mental health.
Time Frame: Baseline-week 12
Population: Monitoring only participants didn't complete week 12, data includes AEs collected as of their last visit
Measure: Mean (Standard Deviation); unit: Number of adverse events
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 2
Number of adverse events | 3 (0) | 4 (0) | 2.5 (2.1)

10. Secondary Outcome: Nicotine Withdrawal Symptoms: Mean Difference (Week 16 - Baseline)
Description: Symptoms will be assessed using the Minnesota Withdrawal Scale (MNWS), a 9-item self-rated scale of nicotine withdrawal symptoms, with scores ranging from 0 - 36, where higher scores indicate a greater degree of withdrawal. The difference between baseline and Week 16 will be computed for each participant.
Time Frame: Baseline to Week 16
Population: Participants in the placebo and monitoring group didn't provide post baseline outcome measure data, and therefore were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 0 | 0
score on a scale | -7 (0) |  |

11. Secondary Outcome: Intensity of Nicotine Craving: Mean Difference (Week 12 - Baseline)
Description: A Visual Analogue Scale was used to measure intensity of nicotine craving. The scale ranged from 0 (no desire at all) to 7 (unable to resist). Higher scores represent more intense nicotine craving.
Time Frame: Baseline to week 12
Population: Measure data was not collected from any enrolled participant.
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Severity of Nicotine Craving: Mean Difference (Week 12 - Baseline)
Description: Severity of nicotine cravings will be assessed using the Questionnaire of Vaping Craving (QVC), a 10-item measure of vaping craving, with scores ranging from 10 - 70, where higher scores indicate greater craving for vaping products. The difference between baseline and Week 12 will be computed for each participant.
Time Frame: Baseline to Week12
Population: participants in the monitoring group didn't provide post baseline outcome measure therefore were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
score on a scale | -16 (0) | -18 (0) |

13. Secondary Outcome: Severity of Clinical Symptoms (Mood and Anxiety): Mean Difference (Week 16 - Baseline)
Description: Severity of clinical symptoms will be assessed by the Mood and Anxiety Symptoms Questionnaire (MASQ-D30), a 30-item measure ranging from 30 - 150, with higher scores indicating a greater degree of clinical distress. The difference between baseline and Week 16 will be computed for each participant.
Time Frame: Baseline-week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo | Monitoring Only
Number analyzed (Participants) | 1 | 1 | 0
score on a scale | -11 (0) | -12 (0) |

14. Other Pre Specified Outcome: Amount of Substances Other Than Nicotine Consumed
Description: Assessed with timeline follow back where individuals report the number of days, times, and amount of alcohol, tobacco, marijuana, and non-medical prescription drugs consumed since last study visit.
Time Frame: Baseline-week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 24 weeks.
Arm/Group | Varenicline | Placebo | Monitoring Only
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=1) | Placebo (N=1) | Monitoring Only (N=2)
Kidney Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=1) | Placebo (N=1) | Monitoring Only (N=2)
Increased Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wisdom Teeth Removal (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Appetite Excessive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04602494/Prot_SAP_000.pdf